CLINICAL TRIAL: NCT05829213
Title: A Modified "Arch-bridge-type" Esophagogastric Reconstruction Method After Laparoscopic Proximal Gastrectomy
Brief Title: A Modified Esophagogastric Reconstruction Method After Laparoscopic Proximal Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, Dr. Prof., Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023YJZ11
Record Dates: First submitted 2023-03-21; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Proximal Gastric Adenocarcinoma; Adenocarcinoma of Esophagogastric Junction; Anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "arch-bridge-type" reconstruction arm (Experimental): In this arm, patients will receive proximal gastrectomy and "arch-bridge-type" reconstruction.
  Interventions: Procedure: "arch-bridge-type" esophagogastric reconstruction after proximal gastrectomy

INTERVENTIONS:
Procedure: "arch-bridge-type" esophagogastric reconstruction after proximal gastrectomy — 1. The lymphadenectomy is performed according to the Japanese Gastric Cancer Treatment Guidelines
  2. Transection of the esophagus is performed using a linear stapler 2cm away from the proximal end of the tumor.
  3. Creating the seromuscular flap ("arch-bridge")
  4. The remnant stomach is then inserted into the abdominal cavity, and pneumoperitoneum is re-established to perform the intracorporeal anastomosis.

SUMMARY:
The double-flap technique (DFT) is an effective digestive tract reconstruction method after proximal gastrectomy (PG) to reduce the incidence of postoperative reflux esophagitis. But its clinical application is restricted due to the technical complexity. Our surgical team devise a modified esophagogastric reconstructive method which we term the "arch-bridge-type" reconstruction based on the principle of DFT. The aim of this single-arm prospective study is to assess the safety and feasibility of the "arch-bridge-type" reconstruction after PG.

DETAILED DESCRIPTION:
1. The lymphadenectomy is performed according to the Japanese Gastric Cancer Treatment Guidelines.
2. Transection of the esophagus is performed using a linear stapler 2cm away from the proximal end of the tumor.
3. Creating the seromuscular flap ("arch-bridge"):

(1) The stomach is resected by a linear stapling device. (2) A "匚" shaped seromuscularflap (3.0cm×4.0cm) is created utilizing electrocautery extracorporeally by dissecting submocosal and muscular layer of the anterior wall of the remnant stomach.

(3) The opening of the flap is interrupted sutured by 4-0 absorbable suture, then the "arch-bridge" is created.

4.The remnant stomach is then inserted into the abdominal cavity, and pneumoperitoneum is re-established to perform the intracorporeal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven proximal gastric cancer or adenocarcinoma of esophagogastric junction
* diameter of the tumor less than 4cm
* ECOG performance status score ≤2
* no distant metastasis
* informed consent is signed

Exclusion Criteria:

* metastatic gastric cancer or metastatic adenocarcinoma of esophagogastric junction
* remnant gastric cancer
* patient requires emergency surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Surgical safety | From surgery day to 30 days after surgery
  The incidence of postoperative complications which were graded using the Clavien-Dindo classification system. The postoperative complications include anastomotic leackage, anastomotic stenosis, abdominal bleeding, gastric emptying disorder, pneumonia complications, etc.
Postoperative long-term quality of life (QoL) | 1 year after surgery
  The QoL is evaluated by postgastrectomy symptom assessment scale (PGSAS-45). Postoperative reflux, abdominal pain, postprandial discomfort, dyspepsia, diarrhea, constipation, dumping syndrome, weight change, food intake per meal, frequency of additional meals, digestive ability, daily work ability, and satisfaction with quality of life will be evaluated in PGSAS-45.

SECONDARY OUTCOMES:
Postoperative body weight status | 1 year after surgery
  Body weight loss will be recorded in outpatient.
Postoperative reflux esophagitis | 1 year after surgery
  Reflux esophagitis will be evaluated by gastroscopy. Reflux esophagitis was graded by the Los Angeles classification.
Refinement of surgery | From surgery day to 30 days after surgery
  During the operation, the whole process of the operation will be videotaped by laparoscopy, and after the operation, the change of the technical process of the operation was judged by comparing the operation in the video and the scheduled operation steps before the operation. In case of technical changes, the surgical team will communicate and discuss with the chief surgeon, and decide whether to adjust and optimize the surgical technique based on the postoperative situation of the patient, so as to form new technical details. Objective metrics include the total operative time, the time of esophagogastric anastomosis, the time of creating the" arch-bridge", intraoperative blood loss, the number of retrieved lymph nodes will be collected.
Postoperative hemoglobin | 1 year after surgery
  Laboratory tests will be done to evaluate the level of hemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, MD PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Ziyu Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No